CLINICAL TRIAL: NCT02274272
Title: Effects of Genmont Probiotic on Improve the Level of Blood Glucose and Other Diabetic Associate Parameter in Type 2 Diabetes Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GenMont Biotech Incorporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P201404-31
Record Dates: First submitted 2014-10-08; First posted 2014-10-24 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Type 2 Diabetes
Keywords: lactobacillus reuteri; type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Placebo Capsules (Placebo Comparator)
  Interventions: Other: placebo
- ADR-1 (Experimental): Lactobacillus reuteri GMNL-89
  Interventions: Other: ADR-1
- GMNL-263 (Experimental): Lactobacillus reuteri GMNL-263
  Interventions: Other: GMNL-263

INTERVENTIONS:
Other: ADR-1 — two ADR-1 capsules, once daily, QD
  Other Names: Lactobacillus reuteri GMNL-89
  Arms: ADR-1
Other: GMNL-263 — two GMNL-263 capsules, once daily, QD
  Other Names: Lactobacillus reuteri GMNL-263
  Arms: GMNL-263
Other: placebo — two placebo capsules, once daily, QD
  Arms: Placebo Capsules

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of probiotics ADR-1/GMNL-263 capsules (Lactobacillus reuteri ADR-1/ Lactobacillus reuteri GMNL-263) for the treatment of adults with type2 DM.

DETAILED DESCRIPTION:
Background：Based on animal studies, intake of probiotic bacteria was suggested to improve insulin sensitivity by reducing inflammation.

Objective ： The objective of this study was to determine the effects of supplementation with the probiotic strain Lactobacillus reuteri ADR-1(ADR-1) and Lactobacillus reuteri GMNL-263 (GMNL-263) over six months on metabolic profiles, intestinal microbiota profiles and biomarkers of inflammation in type 2 diabetes patents. Methods ： This randomized double-blind placebo-controlled clinical trial was performed on 120 diabetic patients. Subjects were divided into 3 groups: 40 subjects in the group A received placebo, 40 subjects in the group B received ADR-1 (4 x 109 colony-forming units/d), and 40 subjects in the group C received GMNL-263. (2 x 1010 cells/d) for 6 months. Fasting blood samples were taken at baseline and after intervention to measure metabolic profiles and biomarkers of inflammation including C reactive protein (CRP), Interleukin 6 (IL-6) and Tumor necrosis factor-alpha( TNF-α). The intestinal microbiota profiles were detected in stool samples by real-time polymerase chain reaction (RT-PCR).

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes with a duration> 6 months
2. 7 % < HbA1c ≦ 10 %
3. Adults 25- 70 years of age
4. BMI>18.5

Exclusion Criteria:

1. Pregnancy
2. Subjects with any other serious diseases such as cancer (patient with benign tumor under medical control should not be ruled out), kidney failure / dialysis, heart disease, stroke.
3. Autoimmune Disease
4. Administration of other healthy food for diabetes 4 weeks before inclusion
5. Administration of probiotic 4 weeks before inclusion
6. Administration of antibiotics 4 weeks before inclusion
7. Participation in other clinical trials
8. ALT/SGPT or AST/SGOT > 3x upper limit of normal (ULN)
9. eGFR<30mL/min/1.73m2
10. Subjects who is lack of physical integrity of gastrointestinal tract, or malabsorption syndrome, or inability to take oral medication.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2014-10; Primary Completion 2017-04 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Change in blood sugar | 6 months
  Fasting blood samples of 120 diabetic patients will be were taken at baseline and after intervention to measure blood sugar(mg/dL) and HbA1c(%).
Change in blood fat | 6 months
  Fasting blood samples of 120 diabetic patients will be were taken at baseline and after intervention to measure cholesterol(mg/dL) ,triglycerides(TG, mg/dl), high density lipoprotein (HDL, mg/dl), low density lipoprotein (LDL, mg/dl).

SECONDARY OUTCOMES:
Change in the DM marker | 6 months
  Fasting blood samples of 120 diabetic patients will be were taken at baseline and after intervention to measure insulin(μIU/mL), C-peptide(ng/mL), Homeostasis model assessment for insulin resistance (HOMA-IR, ratio)

CONTACTS AND LOCATIONS:
Overall Officials: yi shing Chen, PhD, Study Director — GenMont Biothech Incorporation
Locations (1):
- Genmont, Tainan, Taiwan